CLINICAL TRIAL: NCT06784115
Title: A REminder App to Optimize Bladder FILLing in Patients with ProstAte Cancer Receiving HYPO-fractionated Radiotherapy
Acronym: REFILLPAC-HYPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Southern Denmark (Other); University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REFILL-PAC-HYPO
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer Patients Treated by Radiotherapy
Keywords: prostate cancer; radiotherapy; hypofractionation; mobile application; bladder filling
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Support by a reminder app (Experimental): Patients are supported by a Reminder App. The purpose of the app is to remind patients irradiated for prostate cancer in an intuitive, unobtrusive and supportive way to drink 300 ml of water 45 minutes prior to each radiation session. This is supposed to have an impact on the number of bladder volumes <200 ml. Bladder volumes <200 ml were previously shown to be associated with increased urinary toxicity.
  Interventions: Device: Reminder App

INTERVENTIONS:
Device: Reminder App — The purpose of the app is to remind patients irradiated for prostate cancer in an intuitive, unobtrusive and supportive way to drink 300 ml of water 45 minutes prior to each radiation session.

SUMMARY:
The primary goal of this study is to assess the impact of an app that reminds patients treated with hypofractionated radiotherapy (HF-RT) for prostate cancer to drink water prior to each radiotherapy session on the number of bladder volumes <200 ml during the HF-RT course and to demonstrate that this number is lower than without using an app (historical control group).

DETAILED DESCRIPTION:
Prostate cancer is one of the most common solid malignancies worldwide. Many patients receive normo-fractionated (5 × 2.0 Gy per week) external beam radiotherapy (EBRT) alone with 74-80 Gy in 37-40 fractions over 7.5 to 8 weeks Since three randomized trials have demonstrated non-inferiority of moderately hypo-fractionated RT (HF-RT) when compared to normo-fractionated EBRT, the use of HF-RT has become more popular, particularly for patients with low or intermediate prostate cancer. Two of three randomized trials used 20 x 3.0 Gy for HF-RT. Radiotherapy of prostate cancer, irrespective of the type of fractionation, may be associated with significant acute urinary toxicity such as cystitis, particularly if the volume of the urinary bladder is small. Three studies showed that bladder volumes <200 ml or <180 ml, respectively, were associated with increased acute or late urinary toxicity. Therefore, it appears important to achieve bladder volumes >200 ml at as many radiation fractions as possible. In a very recent study of our group that investigated the bladder volumes at each of the 20 fractions in 76 patients receiving HF-RT alone with 20 x 3.0 Gy, the mean and median numbers of radiation fractions with bladder volumes <200 ml were 13.4 (SD, standard deviation = 6.7) and 16.0 (IQR, interquartile range 8.0 - 19.0) fractions, respectively. Whereas in the subgroup of 24 patients with pre-radiotherapy bladder volume of at least 200 ml the mean and median numbers of radiation fractions with bladder volumes <200 ml were only 7.9 (SD = 5.9) and 8.0 (IQR 3.5 - 11.0), respectively, the mean (16.0, SD = 5.5) and median (19.0, IQR 14.5 - 20.0) were significantly higher (p<0.001) in the subgroup of 52 patients with pre-radiotherapy bladder volumes <200 ml. Therefore, there is a medical need for improvement especially in the latter subgroup. Several studies investigated the role of drinking protocols. Patients were asked to drink a certain amount of water prior to the planning computed tomography (CT-simulation) and the radiotherapy sessions. Drinking a certain amount of water at a specific point in time may require considerable discipline from the mainly elderly or very elderly patients. These considerations led to the idea of developing a mobile application (app) that reminds the patients prior to each radiation session to drink a certain amount of water. The present study investigates the number of radiation fractions with bladder volumes <200 ml in a prospective cohort of patients treated with HF-RT using a such a reminder app. In addition, the study evaluates whether the use of the reminder app leads to a significant reduction of the proportion of fractions with bladder volumes <200 ml in patients receiving HF-RT when compared to a historical control group not supported by an app.

Endpoints: The primary endpoint is the number of radiation fractions with bladder volumes <200 ml at the end of radiotherapy. In addition, patient satisfaction with the reminder app and the impact of the reminder app on the use of health technology are evaluated.

General trial design and duration: This is a single-arm prospective study, which will investigate the effect of a reminder app on the number of radiation fractions with bladder volumes <200 ml during a course of HF-RT (20 x 3.0 Gy over 4 weeks) for definitive treatment of prostate cancer in comparison to a historical control group of 52 patients. The historical control group is considered appropriate for the comparison to the cohort of the present study, since all patients of the control group were treated very recently (2022-2024) with HF-RT alone in centers participating in the present study and received a Cone Beam Computed Tomography prior to each radiation fraction, which allowed assessment of the bladder volume as precisely as in the present study.

Recruitment of all 27 patients is planned to be completed within 20 months. The follow-up will end directly after the radiotherapy course, which is scheduled to take 4 weeks. This equals a total running time for the study of 21 months.

In accordance with the previous study assessing the number of fractions with bladder volumes <200 ml during a course of HF-RT for definitive treatment of prostate cancer, the following characteristics will be recorded to allow adequate comparison with the historical control group: Initial (pre-radiotherapy) bladder volume, body-mass index (BMI), age, prostate volume prior to radiotherapy, Karnofsky performance score (KPS), level of prostate-specific antigen (PSA), Gleason score, T-stage, risk group of prostate cancer, and antihormonal therapy.

Sample size calculation: The primary goal of this study is to assess the impact of an app that reminds patients receiving HF-RT for prostate cancer to drink water prior to each radiotherapy session on the number of fractions with bladder volumes <200 ml during the HF-RT course and to demonstrate that this number is lower than without using an app (historical control group). To allow for a skewed distribution of the primary endpoint, the Wilcoxon-Mann-Whitney test will be applied for confirmatory statistical analysis.

In the external historical control group consisting of 52 patients, the mean number of radiation fractions with bladder volumes <200 ml was 16.0 (SD 5.5), and the median number was 19.0 fractions (IQR 14.5 - 20.0). A decrease of this mean value by roughly 30% (to 11.2 fractions) is considered clinically relevant. For illustrative purposes, translating this decrease into a non-parametric effect size framework (assuming for simplicity normal distribution) leads to a probability of roughly 0.27 that the number of fractions <200 ml with the reminder app is larger than without the app. Based on this effect size, a sample size of 24 patients in the prospective trial is required for the comparison with the historical control group to ensure 90% power to reach statistical significance with a two-sided Wilcoxon Mann-Whitney-U-test and a 5% significance level. Assuming that roughly 10% of the enrolled patients will not be eligible for the primary analysis, since they have received less than 20 fractions, a total number of 27 patients should be enrolled in this study.

Statistical considerations: All data recorded in the case report forms describing the study population (demographic and clinical characteristics recorded at baseline), efficacy, safety and quality of life will be analyzed descriptively. Categorical data will be presented in contingency tables with frequencies and percentages and their 95% confidence intervals. Continuous data will be summarized with at least the following: frequency (n), median, quartiles, mean, standard deviation (standard error), minimum and maximum. Number of subjects with protocol deviations during the study and listings describing the deviations will be provided.

In general, chi-square tests will be used to compare percentages in a two-by-two contingency table, replaced by Fisher´s exact test if the expected frequency in at least one cell of the associated table is less than 5. Stratified two-by-two contingency tables will be analyzed using Cochran-Mantel-Haenszel tests. Logistic regression models serve as multivariable methods for binary endpoint data. Comparison of ordinal variables between treatment arms will be performed using the asymptotic Wilcoxon-Mann-Whitney test, replaced by its exact version in case of ordinal categories with small number of categories and/or sparse data within categories. Any shift in location of quantitative variables between study groups will be performed with the Wilcoxon-Mann-Whitney tests as well.

All patients who have started radiotherapy and provide data on the primary endpoint will be analyzed (Full Analysis Set). Data analyses will be performed according to the statistical analysis plan, and which will be finalized prior to database lock and prior to any statistical analysis.

The primary study endpoint is defined as the number of radiation fractions with bladder volumes <200 ml at the end of the HF-RT course (after 20 fractions). Descriptive measures of location and dispersion will be used to describe the results of the prospective study. The impact of patient characteristics on the primary endpoint will be assessed by means of Wilcoxon-two sample tests. These factors include age (<75 vs. ≥75 years), Karnofsky performance score (70-80 vs. 90-100), body-mass index (<30 vs. ≥30=obesity), prostate volume prior to HF-RT (<60 vs. ≥60 mL), PSA-level prior to HF-RT (<10 vs. ≥10 ng/mL), Gleason score (≤7 vs. 8-9), primary tumor stage (T1 vs. T2 or T3), risk group of prostate cancer (low to intermediate vs. high), and antihormonal therapy prior to and/or during the course of HF-RT (no vs. yes).

For confirmatory analysis, the prospective study will be compared with the historical control group by means of a two-sided Wilcoxon-Mann-Whitney two sample test and significance level of 5%. A high degree of comparability of patient population is expected between the prospective trial data and the retrospective patient data set. However, potential heterogeneity of study populations will be identified by comparing the patient characteristics listed above with Wilcoxon-Mann-Whitney tests. Homogeneity is assumed if all resulting p-values are above 20%. Any factor indicating a tendency towards heterogeneity (i.e. p<0.20) will be included in a multivariable count data Poisson regression model with the number of radiation fractions with bladder volumes < 200 ml as dependent variable and including the respective factors and the binary factor (prospective study vs historical control) as independent variables. In case of evidence of overdispersion the Poisson model will be replaced by a negative binomial model.

In addition to the primary study endpoint, secondary endpoints will be subjected to statistical analysis. Since no comparison with historical data is possible, these analyses focus on descriptive statistical analysis only. The results of patient satisfaction will be used to decide whether the app needs modification: In case of a dissatisfaction rate >20%, the reminder app needs modifications. In case of a dissatisfaction rate >40%, it will be considered not useful.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven prostate cancer
2. Indication for definitive HF-RT
3. Possession of and ability to use a smartphone
4. Bladder volume at CT-simulation <200 ml
5. Male gender
6. Age ≥18 years
7. Written informed consent
8. Capacity of the patient to contract

Exclusion Criteria:

1. Radiotherapy of pelvic lymph nodes
2. Expected non-compliance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of fractions with bladder volumes <200 ml at the end of the radiotherapy course | through study completion, an average of 4 weeks
  The primary endpoint is the number of radiation fractions with bladder volumes <200 ml at the end of the radiotherapy course. The bladder volume at each radiation fraction is calculated from the corresponding Cone-Beam Computed Tomography (CBCT).

SECONDARY OUTCOMES:
Rate of patient satisfaction with the reminder app | through study completion, an average of 4 weeks
  Patient satisfaction with the reminder app will be assessed with a specific questionnaire.
Degree of the impact of the reminder app | through study completion, an average of 4 weeks
  The impact of the reminder app on the use of health technology will be assessed with a specific questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr., Principal Investigator — Department of Radiation Oncology, University of Lubeck, Germany
Locations (4):
- Department of Oncology, Vejle Hospital, University Hospital of Southern Denmark, Vejle, Southern Denmark, Denmark
- Germany (2):
  - Medical Practice for Radiotherapy and Radiation Oncology, Hanover, Lower Saxony
  - Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Lübeck, Schleswig-Holstein
- Radiation Oncology Department, Hospital Universitario Cruces/Biobizkaia Health Research Institute University of the Basque Country, Barakaldo, Basque Country, Spain

IPD SHARING:
Plan to Share IPD: No